CLINICAL TRIAL: NCT01492179
Title: A Comparison Between Continuous Infusion vs. Patient Controlled Intraabdominal Injection of Local Anesthetics for Treatment of Postoperative Pain After Abdominal Hysterectomy. A Randomized, Double-blind Study.
Brief Title: Intravenous or Intra-abdominal Local Anesthetics for Postoperative Pain Management.
Acronym: PoPuLAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Anil Gupta, Associate Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20111212
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Uterine Myoma; Persistent Post-menpausal Bleeding; Uterine Cancer
Keywords: Surgery: Abdominal hysterectomy; Anesthetics: Local; Postoperative: Pain; Drugs: Morphine
MeSH Terms: conditions — Myofibroma; Uterine Neoplasms; Pain, Postoperative | interventions — Saline Solution; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous Lidocaine (Active Comparator): Intravenous lidocaine would be administered as an infusion for pain management both intra- and post-operatively.
  Interventions: Drug: Intravenous Lidocaine
- Intra-abdominal Lidocaine (Active Comparator): Lidocaine would be administered intermittently, once each hour intra-abdominally for postoperative pain management.
  Interventions: Drug: Intra-abdominal Lidocaine
- Normal saline (Placebo Comparator): Normal saline would be administered intra-abdominally and intravenously in the same patient. Rescue analgesia in the form of morphine (PCA) would be used for pain management.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Normal saline — Normal saline would be administered intravenously and intra-abdominally.
  Arms: Normal saline
Drug: Intravenous Lidocaine — Standardized infusion of lidocaine during 24 h. 100 mg bolus and 50 mg/h during 24 h would be administered.
  Other Names: Xylocaine 5 mg/ml
  Arms: Intravenous Lidocaine
Drug: Intra-abdominal Lidocaine — Lidocaine 5 mg/ml; 100 mg would be administered intraoperatively intra-abdominally and subsequently 50 mg/h as intermittent injection intra-abdominally during 24 h
  Other Names: Xylocaine 5 mg/ml
  Arms: Intra-abdominal Lidocaine

SUMMARY:
Local anesthetics (LA) are increasingly used for postoperative pain management. Speicifically, several studies have found benefit of LA injected intra-abdominally following abdominal hysterectomy. However, it remains unclear whether the pain relief seen is due to local anesthetic mechanisms within the abdominal cavity or through systemic absorption. The aim of this study is to assess whether lidocaine administered intravenously has similar analgesic efficacy as the same dose administered intra-abdominally in patients undergoing abdominal hysterectomy. All patients would have rescue analgesia using the patient controlled analgesia (PCA) pump with morphine in order to achieve adequate pain management during 24 h.

DETAILED DESCRIPTION:
Abdominal hysterectomy with or without salipingo-oophorectomy is associated with moderate-severe postoperative pain. Poor pain control in the postoperative period can lead to increased postoperative morbidities and poor quality of life. Furthermore, an emerging clinical literature suggests that acute pain may rapidly evolve into chronic pain if poorly treated. A meta-analysis of the literature found that > 30% patients had chronic pain one year after abdominal hysterectomy (5). Therefore, efficient postoperative pain management is imperative for the patient and is one of the new pain management standards recommended recently.

Local anesthetics (LA) have been infiltrated subcutaneously, infused intra-abdominally, as well as injected into the peritoneal cavity as a single dose at the end of the operation following abdominal hysterectomy with variable effects. When injected as a single dose, analgesia is limited to approximately 2-4 hours due to the short duration of action of local anesthetics. In one recent study, the authors used a catheter inserted intra-abdominally and local anesthetic or placebo infusion into the abdominal cavity for 24 h postoperatively and found a reduction in postoperative analgesic requirements by 40% during 4-24 h. In another study, the investigators found that LA injected intermittently intra-abdominally resulted in better pain relief compared to intra-abdominal infusions.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* 30 - 75 yrs
* Informed consent
* 50 - 100 kg

Exclusion Criteria:

* Allergy to LA
* Chronic pain
* Major liver/kidney insufficiency
* AV Block 1-2 Participation in another clinical trial

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 0 - 24 h postoperatively
  Total rescue morphine consumption during 0 - 24 h would be the primary endpoint

SECONDARY OUTCOMES:
Postoperative pain | 4 h postoperatively
  Postoperative pain measured on the numeric rating scale (0 - 10) would be measured at 4 h
Plasma concentration of lidocaine | 24 h
  The plasma concentration of LA lidocaine would be analysed at 24 h in order to assess whether the LA absorption from the abdomen is similar to that administered intravenously.
Length of Hospital stay | 1-5 days
  The time to discharge home would be assessed using standardized criteria for home discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Axelsson, MD, PhD, Study Director — Örebro University Hospital, Örebro, Sweden
Locations (1):
- Örebro University Hospital, Örebro, Sweden